CLINICAL TRIAL: NCT01984593
Title: Impact of Yoga on Blood Pressure, Quality of Life and Stress in Patients With Hypertension - A Randomized Controlled Multicenter Trial in Primary Care
Brief Title: Impact of Yoga on Blood Pressure, Quality of Life and Stress in Patients With Hypertension
Acronym: YHIP2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: The Swedish Research Council (Other Government)
Responsible Party: Principal Investigator, Moa Wolff, General Practitioner, Region Skane
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Region Skane
Record Dates: First submitted 2013-11-08; First posted 2013-11-14 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-11

CONDITIONS: Hypertension
Keywords: Yoga; Hypertension; Quality of Life; Primary Health Care; Stress; Anxiety; Depression
MeSH Terms: conditions — Hypertension; Anxiety Disorders; Depression | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): No changes will be made for the participants in the control group, but they will undergo the same measurements and evaluations as the intervention group.
- yoga (Active Comparator): Two yoga exercises to perform at home 15 minutes twice daily.
  Interventions: Other: Yoga

INTERVENTIONS:
Other: Yoga — The participants in the Yoga group will get a private doctors appointment (20 minutes) where they get instructions for two yoga exercises to perform at home 15 minutes twice a day.
  The two yoga exercises were:
  1. "Left nostril breathing" - deep breaths in and out through the left nostril while sitting or lying down, with the right nostril closed off by the right thumb or an earplug (about 11 minutes); and
  2. "Spinal flex" - movement that alternates between flexing the spine forwards (arching) and relaxing the spine back in time with deep breaths while sitting in a chair (about 4 minutes).
  Arms: yoga

SUMMARY:
The purpose of this study is to determine the effects of a short yoga program practiced daily at home on blood pressure, quality of Life and stress. The subjects of the study are primary health care patients diagnosed with hypertension, with or without current medication.

DETAILED DESCRIPTION:
Hypertension is one of the most common diseases in the world, affecting approximately 26% of the adult population. Persistent hypertension increases the risk of developing coronary heart disease, stroke and other cardiovascular diseases, such as heart failure. Hypertension is a common diagnosis in primary health care and the societal costs of examination and treatment of hypertension and its consequences are considerable.

The YHIP-study (The Impact of Yoga on Blood Pressure and Quality of Life in Patients With Hypertension), that investigated yoga as additional treatment for hypertension on primary care patients, showed that a short yoga program practiced daily at home had a blood pressure lowering effect as well as a positive effect on self-rated quality of life compared to control.

Other previous studies have demonstrated positive effects of yoga on blood pressure, quality of life, subjective well-being and stress. However, these studies are relatively few and we need to further investigate the possibility of using yoga as a treatment in primary health care.

If the yoga intervention shows to be effective, yoga exercises may be useful as a supplementary BP therapy in addition to medical treatment when prescribed by primary care physicians. It is to be hoped that patients will also experience a higher quality of life and less stress if they perform yoga on a regular basis.

ELIGIBILITY:
Inclusion Criteria:

* 30-80 years old
* Diagnosed with hypertension since at least one year
* Blood pressure 130-160 mm Hg systolic and/or 85-100 diastolic at the last blood pressure control by doctor or nurse.
* Blood pressure within inclusion- and exclusion-limits at baseline control

Exclusion Criteria:

* Blood pressure outside the range of 120-180 systolic and 80-110 diastolic at the last blood pressure control or at baseline control.
* Medical adjustments regarding hypertension within 4 weeks prior to begin of study.
* Expected inability to understand instructions about yoga exercises (e.g dementia and mental retardation) or physical or psychical inability to carry out yoga exercises (e.g severe physical or psychical handicap).
* Need for interpreter. Linguistic/language difficulties

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2013-11; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Hypertension | 12 weeks
  At the beginning of the study, all subjects will undergo a standardized blood pressure test with an hypertension monitor. After 12 weeks, all subjects in the intervention and control groups will again be requested to attend a blood pressure testing session

SECONDARY OUTCOMES:
Quality of life | 12 weeks
  At the beginning of the study, all subjects will be requested to fill in a questionnaire about their quality of life (WHOQOL-BREF). After 12 weeks all subjects in the intervention and control groups will fill in the quality of life-form for a second time.

OTHER OUTCOMES:
Stress | 12 weeks
  At the beginning of the study, all subjects will be requested to fill in a questionnaire about their self-rated stress(PSS). After 12 weeks all subjects in the intervention and control groups will fill in the stress-questionnaire once again.
Anxiety and depression | 12 weeks
  At the beginning of the study, all subjects will be requested to fill in a questionnaire with questions regarding anxiety and depression(HAD). After 12 weeks all subjects in the intervention and control groups will complete the questionnaire once again.

CONTACTS AND LOCATIONS:
Overall Officials: Moa Wolff, MD, Principal Investigator — Center for Primary Health Care Research, Lunds University
Locations (1):
- Center for Primary Health Care Research, Lunds University, Malmo, Sweden